CLINICAL TRIAL: NCT03667872
Title: Efficacy and Safety of MRI Compatible and Long-term LFP Recordable Deep Brain Stimulation in Patients With Treatment-Resistant Depression
Brief Title: Efficacy and Safety of DBS in Patients With Treatment-Resistant Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Pins Medical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PINS-029
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Last update posted 2018-12-27 (Actual); Status verified 2018-12

CONDITIONS: Treatment Resistant Depressive Disorder
Keywords: Deep Brain Stimulation; Habenula; Functional magnetic resonance imaging
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Device (Experimental): MRI compatible and LFP recordable implantable stimulator
  Interventions: Procedure: Bilateral implantation of DBS system to Habeluna

INTERVENTIONS:
Procedure: Bilateral implantation of DBS system to Habeluna — Bilateral implantation of MRI compatible and LFP recordable DBS system to Habeluna

SUMMARY:
The habenula (Hb) is an ancient structure, located at the center of the dorsal diencephalic conduction system, a pathway involved in linking forebrain to midbrain regions. An increasing number of studies indicated that the lateral habeluna (LHb) is overactivity during depressive behaviors in rats, where it could drive the changes in midbrain monoamine neurotransmitter linked to depression. However, the efficiency and mechanism of deep brain stimulation (DBS) of the LHb and/or its major afferent bundle (i.e., stria medullaris thalami) could treat treatment-resistant major depression (TRD) is still unclear. This research will investigate the effectiveness and mechanism of bilateral MRI Compatible and Long-term LFP Recordable DBS to habenula and/or its major afferent bundle for treatment TRD patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years old;
* DSM-IV diagnosis of Major depression disorder of psychiatrists;
* More than 3 year's history of depression and failure to respond to a minimum of three different antidepressant treatments;
* Failure or intolerance or unwilling of an adequate course of electroconvulsive therapy (ECT) during any episode;
* HAMD-17≥20;
* GAF≤50；
* Capacity to provide informed consent (understanding of the study purpose and methods);

Exclusion Criteria:

* Obvious medical and psychiatric comorbidities;
* Alcohol or substance abuse/dependence within 12 months;
* Antisocial personality disorder, dementia, current tic disorder;
* Subject has a history of 2 or more suicide attempts < 12 months prior to the screening testing;
* Pregnancy and/or lactation;
* There are contraindications for DBS surgery and chronic stimulation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2019-01-15 (Estimated); Primary Completion 2020-06-18 (Estimated); Study Completion 2022-06-18 (Estimated)

PRIMARY OUTCOMES:
Change in the Hamilton Anxiety Scale | Baseline（preoperative）,3 months, 6 months, 12months
  Change in the Hamilton Anxiety Scale after the DBS on

CONTACTS AND LOCATIONS:
Locations (1):
- Habenula DBS, Shenzhen, Shenzhen, China